CLINICAL TRIAL: NCT03608735
Title: Prevalence of Functional Gastrointestinal Disorders (FGIDs) and Related Signs and Symptoms in Infants and Toddlers in Thailand
Brief Title: Prevalence of Functional Gastrointestinal Disorders (FGIDs), Related Signs and Symptoms in Infants/Toddlers in Thailand
Acronym: GI_Planet
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: ObvioHealth (Industry)
Responsible Party: Sponsor
Other Study IDs: EBB17GC17070_1 / OBVIO-DAN-004
Record Dates: First submitted 2018-07-17; First posted 2018-08-01 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevalence and impact of Functional Gastrointestinal Disorders (FGIDs) and Related Signs and Symptoms in Infants and Toddlers in Thailand

DETAILED DESCRIPTION:
Primary:

To assess the prevalence of specific FGIDs (infant regurgitation, infantile colic and functional constipation) and related signs and symptoms in infants and toddlers in Thailand, according to information provided by the parents.

Secondary:

To assess the impact of FGIDs (Infant regurgitation, Infantile colic and functional constipation) and related signs and symptoms of infants and toddlers on the quality of life (QoL) of parents/caretakers and family, according to information provided by the parents.

Exploratory:

To assess treatments and practices employed in real-life to manage FGIDs according to the Rome IV criteria (infant regurgitation, infantile colic, and functional constipation) and related signs and symptoms in infants and toddlers, according to information provided by the parents.

ELIGIBILITY:
Inclusion Criteria:

1. Parent of otherwise healthy infants and/or toddlers from one of the age groups: 3±1 months, 6±1 months, 9±1 months, 12±1 months, or 18±1 months
2. Parent answering the online survey questionnaire attends to the child more than 50% of the time
3. Informed consent from one or both parents (according to local laws) and/or legal guardian.
4. Parent should have reliable access to the internet and a reliable device such as a computer, tablet or smartphone to complete the online survey questionnaire

Exclusion Criteria:

1. Parent who is not adequately comfortable in the language in which the online survey questionnaire will be completed
2. Inability of the parent to answer the survey questionnaire online.
3. Infants and Toddlers who underwent surgery under general anesthesia

Ages: 2 Months to 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: otherwise healthy infants and toddlers aged 2 to 19 months
Sampling Method: Non-Probability Sample
Enrollment: 7908 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
To determine the ROME IV Criteria score | 1 day
  FGIDs according to the ROME IV criteria (infant regurgitation, infantile colic, and functional constipation), related signs and symptoms in infants and toddlers based on parent's response in the survey questionnaires. Scale measures 1-7

SECONDARY OUTCOMES:
To measure Quality of Life using modified Pediatric Quality of Life Inventory™ | 1 day
  Pediatric Quality of Life Inventory of the parents/caretakers and the family (using modified PedsQL™ Family Impact Module, Scale 0 -144)

OTHER OUTCOMES:
To determine use of medication for the management of FGID via Adapted Parent Report Form for Infants and Toddlers Questionnaire on Paediatric Gastrointestinal Symptoms, Rome IV (R4PDQ-toddler) | 1 day
  Use of medications for FGIDs and related signs and symptoms Use of treatments (other than medications or nutritional supplements) for FGIDs and related signs and symptoms Use of nutritional supplements for FGIDs and related signs and symptoms Use of other remedies for FGIDs and related signs and symptoms Visit to doctor, healthcare professional, clinic, and/or hospital for FGIDs and related signs and symptoms
To determine use of treatment for the management of FGID via Adapted Parent Report Form for Infants and Toddlers Questionnaire on Paediatric Gastrointestinal Symptoms, Rome IV (R4PDQ-toddler) | 1 day
  Use of treatment (other than medication) for FGIDs and related signs and symptoms Use of treatments (other than medications or nutritional supplements) for FGIDs and related signs and symptoms Use of nutritional supplements for FGIDs and related signs and symptoms Use of other remedies for FGIDs and related signs and symptoms Visit to doctor, healthcare professional, clinic, and/or hospital for FGIDs and related signs and symptoms
To determine use of nutritional supplements for the management of FGID via Adapted Parent Report Form for Infants and Toddlers Questionnaire on Paediatric Gastrointestinal Symptoms, Rome IV (R4PDQ-toddler) | 1 day
  Use of supplements for FGIDs and related signs and symptoms Use of treatments (other than medications or nutritional supplements) for FGIDs and related signs and symptoms Use of nutritional supplements for FGIDs and related signs and symptoms Use of other remedies for FGIDs and related signs and symptoms Visit to doctor, healthcare professional, clinic, and/or hospital for FGIDs and related signs and symptoms
To determine use of other remedies for the management of FGID via Adapted Parent Report Form for Infants and Toddlers Questionnaire on Paediatric Gastrointestinal Symptoms, Rome IV (R4PDQ-toddler) | 1 day
  Use of other remedies (other than medication, supplements) for FGIDs and related signs and symptoms Use of treatments (other than medications or nutritional supplements) for FGIDs and related signs and symptoms Use of nutritional supplements for FGIDs and related signs and symptoms Use of other remedies for FGIDs and related signs and symptoms Visit to doctor, healthcare professional, clinic, and/or hospital for FGIDs and related signs and symptoms
Visit to doctor, healthcare professional, clinic, and/or hospital for FGIDs and related signs and symptoms via Adapted Parent Report Form for Infants and Toddlers Questionnaire on Paediatric Gastrointestinal Symptoms, Rome IV (R4PDQ-toddler) | 1 day
  Visit to doctor, healthcare professional, clinic, and/or hospital for FGIDs and related signs and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Busara Charoenwat, MBBS, Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand